CLINICAL TRIAL: NCT00768703
Title: Percutaneous Endoscopic Tracheal Plug/Unplug for Congenital Diaphragmatic Hernia
Brief Title: Percutaneous Endoscopic Tracheal Plug/Unplug for CDH (Congenital Diaphragmatic Hernia)
Status: No longer available | Type: Expanded Access
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Hanmin Lee, Principal Investigator, University of California, San Francisco
Other Study IDs: 10-01765; TO CDH (Other: UCSF(University of California, San Francisco) Fetal Treatment Center)
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Severe Congenital Diaphragmatic Hernia
Keywords: Congenital diaphragmatic hernia; lung-head ratio; percutaneous tracheal occlusion; fetal intervention
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Device: Percutaneous endoscopic fetal tracheal occlusion/unocclusion — Between 26-28 wks' gestation, percutaneous endoscopic placement of the tracheal balloon. Between 32-34 wks' gestation, percutaneous endoscopic removal of the balloon.
  Other Names: Goldvalve Balloon and MiniTorquer Delivery Microcatheter

SUMMARY:
Congenital diaphragmatic hernia is an anatomically simple birth defect in which contents of the fetal abdomen migrate into the chest due to incomplete formation of the diaphragm. Herniation of viscera into the chest prevents the fetal lungs from developing and growing to normal size. In the most severe cases, there is significant morbidity and mortality at birth. For these fetuses, fetal intervention may improve outcomes by enabling the lungs to grow enough in utero that they are capable of sustaining life after birth. This unblinded, non-randomized trial will assess the safety and efficacy of the use of the Goldvalve balloon and MiniTorquer microcatheter to perform percutaneous temporary tracheal occlusion to treat severe CDH in utero. The primary outcome variable will be fetal lung growth due to successful 'plugging/unplugging' of the trachea, as determined by serial lung-head ratio (LHR) measurements. Secondary outcome variables include maternal, fetal and neonatal variables, specifically neonatal survival at 90 days of life. For infants who survive beyond 90 days post-delivery, their families will be offered follow-up (up to 2 years of age and possibly beyond) in the Long-term Infant-to-Adult Follow-up Evaluation (LIFE) Clinic at UCSF.

ELIGIBILITY:
General subject population: Pregnant women in the second trimester, at least 18 years of age, and of any and all ethnic backgrounds.

Inclusion Criteria:

* Confirmed diagnosis of CDH
* Normal fetal echocardiogram
* Normal karyotype
* Fetal liver herniated into the left hemithorax
* Lung-head ratio (LHR) is 1.0 or less, calculated between 24-26 weeks' gestation
* Fetus is between 26 and 28 weeks' gestation
* Singleton pregnancy
* Mother meets psychosocial criteria
* Pre-authorization from third-party payor for fetal intervention, or ability to self-pay.

Exclusion Criteria:

* Failure to meet all inclusion criteria
* Other congenital anomalies detected on ultrasound
* Contraindication to abdominal surgery or general anesthesia
* Allergy to latex
* Preterm labor, preeclampsia, or uterine anomaly (e.g., large fibroid tumor)
* Family unable or refuses to stay in San Francisco for duration of the tracheal occlusion period and for the duration of the pregnancy as medically necessary.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Lee, MD, Principal Investigator — University of California, San Francisco Fetal Treatment Center
Locations (1):
- University of California, San Francisco Fetal Treatment Center, San Francisco, California, United States

REFERENCES:
- [Background] Jani JC, Nicolaides KH, Gratacos E, Vandecruys H, Deprest JA; FETO Task Group. Fetal lung-to-head ratio in the prediction of survival in severe left-sided diaphragmatic hernia treated by fetal endoscopic tracheal occlusion (FETO). Am J Obstet Gynecol. 2006 Dec;195(6):1646-50. doi: 10.1016/j.ajog.2006.04.004. Epub 2006 Jun 12. PMID 16769018
- [Background] Done E, Gucciardo L, Van Mieghem T, Jani J, Cannie M, Van Schoubroeck D, Devlieger R, Catte LD, Klaritsch P, Mayer S, Beck V, Debeer A, Gratacos E, Nicolaides K, Deprest J. Prenatal diagnosis, prediction of outcome and in utero therapy of isolated congenital diaphragmatic hernia. Prenat Diagn. 2008 Jul;28(7):581-91. doi: 10.1002/pd.2033. PMID 18634116
- [Background] Cortes RA, Keller RL, Townsend T, Harrison MR, Farmer DL, Lee H, Piecuch RE, Leonard CH, Hetherton M, Bisgaard R, Nobuhara KK. Survival of severe congenital diaphragmatic hernia has morbid consequences. J Pediatr Surg. 2005 Jan;40(1):36-45; discussion 45-6. doi: 10.1016/j.jpedsurg.2004.09.037. PMID 15868556
- [Background] Keller RL, Hawgood S, Neuhaus JM, Farmer DL, Lee H, Albanese CT, Harrison MR, Kitterman JA. Infant pulmonary function in a randomized trial of fetal tracheal occlusion for severe congenital diaphragmatic hernia. Pediatr Res. 2004 Nov;56(5):818-25. doi: 10.1203/01.PDR.0000141518.19721.D7. Epub 2004 Aug 19. PMID 15319458
- [Background] Harrison MR, Keller RL, Hawgood SB, Kitterman JA, Sandberg PL, Farmer DL, Lee H, Filly RA, Farrell JA, Albanese CT. A randomized trial of fetal endoscopic tracheal occlusion for severe fetal congenital diaphragmatic hernia. N Engl J Med. 2003 Nov 13;349(20):1916-24. doi: 10.1056/NEJMoa035005. PMID 14614166
- [Background] Harrison MR, Albanese CT, Hawgood SB, Farmer DL, Farrell JA, Sandberg PL, Filly RA. Fetoscopic temporary tracheal occlusion by means of detachable balloon for congenital diaphragmatic hernia. Am J Obstet Gynecol. 2001 Sep;185(3):730-3. doi: 10.1067/mob.2001.117344. PMID 11568805
- [Background] Ruano R, Ali RA, Patel P, Cass D, Olutoye O, Belfort MA. Fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia: indications, outcomes, and future directions. Obstet Gynecol Surv. 2014 Mar;69(3):147-58. doi: 10.1097/OGX.0000000000000045. PMID 25102346
- [Background] Done E, Gratacos E, Nicolaides KH, Allegaert K, Valencia C, Castanon M, Martinez JM, Jani J, Van Mieghem T, Greenough A, Gomez O, Lewi P, Deprest J. Predictors of neonatal morbidity in fetuses with severe isolated congenital diaphragmatic hernia undergoing fetoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2013 Jul;42(1):77-83. doi: 10.1002/uog.12445. PMID 23444265
- See also: UCSF Fetal Treatment Center — http://fetus.ucsfmedicalcenter.org/